CLINICAL TRIAL: NCT05838716
Title: High-dose Vitamin D Supplementation for ADT-Induced Bone Loss in Older Prostate Cancer Patients
Brief Title: Vitamin D for Prostate Endocrine Therapy
Acronym: ViPER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Luke Peppone, URCC Study Chair, University of Rochester NCORP Research Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: URCC-22053; NCI-2022-07664 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC-22053 (Other: University of Rochester NCORP Research Base); URCC-22053 (Other: DCP); URCC-22053 (Other: CTEP); R01CA258349 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Cholecalciferol; Vitamin D; Absorptiometry, Photon; Bone Density

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (HDVD) (Experimental): Patients receive HDVD PO QW for 52 weeks. Patients also undergo collection of blood and DXA scan on study.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: D Vitamin; Procedure: Dual X-ray Absorptiometry; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QW for 52 weeks. Patients also undergo collection of blood and DXA scan on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Dual X-ray Absorptiometry; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Dietary Supplement: D Vitamin — Given PO
  Other Names: 3-[2-[7a-methyl-1-(1,4,5-trimethylhex-2-enyl)-1,2,3,3a,5,6,7,7a-octahydroinden-4-ylidene]ethylidene]-4-methylidene-cyclohexan-1-ol; Vitamin D; Vitamin D Compound; Vitamin-D
  Arms: Arm I (HDVD)
Procedure: Dual X-ray Absorptiometry — Undergo DXA scan
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA (Bone Density); DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial tests whether high-dose vitamin D works in treating androgen-deprivation therapy (ADT)-induced bone loss in patients with prostate cancer who are undergoing androgen-deprivation therapy. Vitamins are substances that the body needs to grow and develop normally. Vitamin D helps the body absorb calcium. Calcium is one of the main building blocks of bone. A lack of vitamin D can lead to bone diseases such as osteoporosis or rickets. This trial may help researchers determine if high-dose vitamin D helps keep bones strong, lowers number of falls, and lessens fatigue in men getting androgen-deprivation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of high-dose vitamin D (HDVD) supplementation in prostate cancer patients on ADT-induced bone mineral density loss in the total hip over 52 weeks as measured by dual-energy x-ray absorptiometry (DXA).

II. To evaluate the effect of HDVD supplementation in prostate cancer patients on ADT-induced bone mineral density loss in the femoral neck, distal radius, and lumbar spine (L1-L4) over 52 weeks as measured by DXA.

SECONDARY OBJECTIVES:

I. To evaluate the effect of HDVD supplementation on falls over 52 weeks as measured by the Falls History questionnaire.

II. To evaluate the effect of HDVD supplementation on fractures over 52 weeks as determined by the Clinical Record Information - Follow-up Form.

III. To evaluate the effect of HDVD supplementation on quality of life over 52 weeks as measured by the Functional Assessment of Cancer Therapy- Prostate (FACT-P).

EXPLORATORY OBJECTIVE:

I. To evaluate the effect of HDVD supplementation on pain, fatigue, sleep, and activities of daily living over 52 weeks as measured by patient-reported outcomes.

OUTLINE: After undergoing collection of blood and DXA scan, patients are randomized to 1 of 2 arms.

ARM I: Patients receive HDVD orally (PO) once a week (QW) for 52 weeks. Patients also undergo collection of blood and DXA scan on study.

ARM II: Patients receive placebo PO QW for 52 weeks. Patients also undergo collection of blood and DXA scan on study.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with Stage I-IV prostate cancer without metastases to bone (lymph node involvement and prior diagnosis of a primary cancer is allowed)
* Be age 50 years or older
* Be starting ADT or have received their first ADT treatment in the past 6 months, with a total of at least 6 planned months of treatment (both luteinizing hormone-releasing hormone [LHRH] antagonists and LHRH agonists are permitted)
* Have a total serum vitamin D between 10 and 32 ng/ml
* Have a total serum calcium of less than or equal to 10.5 mg/dl
* Have a normal GFR (glomerular filtration rate > 30ml)
* Agree not to take calcium and/or vitamin D supplements for the duration of the intervention other than those provided by the study
* Be able to provide written informed consent
* Be able to swallow pills and capsules
* Be able to speak and read English

Exclusion Criteria:

* Have long term (greater than 3 months) use of any pharmacologic bone-modifying agent including but not limited to oral or intravenous (IV) bisphosphonates, denosumab, or teriparatide prior to enrollment
* Have a diagnosis of stage IV chronic kidney disease
* Have a diagnosis of grade II or greater hypercalcemia (serum calcium greater than 11.5 mg/dl)
* Have a history of hypercalcemia or vitamin D toxicity/sensitivity

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2029-04-29 (Estimated); Study Completion 2029-04-29 (Estimated)

PRIMARY OUTCOMES:
Reduction of bone mineral density (BMD) loss as measured at the total hip | At 52 weeks
  Will determine the efficacy of high-dose vitamin D (HDVD) supplementation versus placebo in reducing BMD loss as measured at the total hip via dual-energy x-ray absorptiometry (DXA) at 52 weeks. Will use analysis of covariance (ANCOVA) with group (vitamin D or placebo) as the main factor, baseline timepoint ([T]1) BMD as covariate, and week 52 (T3) BMD as the outcome. Study site will be included as a random effect independent of residual error. An initial linear mixed model (LMM) will be fit using Restricted Maximum Likelihood (REML) estimation. The significance of the variance due to study site will be tested using the Wald Test.
Reduction of BMD loss as measured at the femoral neck | At 52 weeks
  Will determine the efficacy of HDVD supplementation versus placebo in reducing BMD loss as measured at the femoral neck via DXA at 52 weeks. Will use ANCOVA with group (vitamin D or placebo) as the main factor, baseline (T1) BMD as covariate, and week 52 (T3) BMD as the outcome. Study site will be included as a random effect independent of residual error. An initial LMM will be fit using REML estimation. The significance of the variance due to study site will be tested using the Wald Test.
Reduction of BMD loss as measured at the distal radius | At 52 weeks
  Will determine the efficacy of HDVD supplementation versus placebo in reducing BMD loss as measured at the distal radius via DXA at 52 weeks. Will use ANCOVA with group (vitamin D or placebo) as the main factor, baseline (T1) BMD as covariate, and week 52 (T3) BMD as the outcome. Study site will be included as a random effect independent of residual error. An initial LMM will be fit using REML estimation. The significance of the variance due to study site will be tested using the Wald Test.
Reduction of BMD loss as measured at the lumbar spine | At 52 weeks
  Will determine the efficacy of HDVD supplementation versus placebo in reducing BMD loss as measured at the lumbar spine via DXA at 52 weeks. Will use ANCOVA with group (vitamin D or placebo) as the main factor, baseline (T1) BMD as covariate, and week 52 (T3) BMD as the outcome. Study site will be included as a random effect independent of residual error. An initial LMM will be fit using REML estimation. The significance of the variance due to study site will be tested using the Wald Test.

SECONDARY OUTCOMES:
Change in falls | Baseline up to 52 weeks
  Will use generalized linear mixed models. Logistic regression models will be used to estimate the between group difference in (1) the proportion of participants who experience a fall/fracture (YES/NO) from T1 to T3. Will evaluate the distribution of total number of falls/fractures by Poisson models analysis to estimate the between group difference in (2) the total number of falls/fractures from T1 to T3. Both models (1, 2) will contain group as fixed effect and site as a random effect. Additional adjustment covariates will include falls in the previous 6 months, fractures in the previous 5 years, androgen-deprivation therapy (ADT) dose and duration, stage, radiation therapy, prior surgery, baseline vitamin D, age, body mass index (BMI), and race. Nonsignificant (P > 0.05) covariates will be removed from the model. Will report the estimates and associated 95% confidence intervals as (1) relative risk or (2) rate ratio.
Change in fractures | Baseline up to 52 weeks
  Will use generalized linear mixed models. Logistic regression models will be used to estimate the between group difference in (1) the proportion of participants who experience a fall/fracture (YES/NO) from T1 to T3. Will evaluate the distribution of total number of falls/fractures by Poisson models analysis to estimate the between group difference in (2) the total number of falls/fractures from T1 to T3. Both models (1, 2) will contain group as fixed effect and site as a random effect. Additional adjustment covariates will include falls in the previous 6 months, fractures in the previous 5 years, ADT dose and duration, stage, radiation therapy, prior surgery, baseline vitamin D, age, BMI, and race. Nonsignificant (P > 0.05) covariates will be removed from the model. Will report the estimates and associated 95% confidence intervals as (1) relative risk or (2) rate ratio.
Change in quality of life | Baseline up to 52 weeks
  Will be evaluated by Functional Assessment of Cancer Therapy-Prostate Trial Outcome Index score.

CONTACTS AND LOCATIONS:
Overall Officials: Luke J Peppone, Principal Investigator — University of Rochester NCORP Research Base
Locations (51):
- United States (51):
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Nash UNC HealthCare, Rocky Mount, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Regional Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin